CLINICAL TRIAL: NCT05747170
Title: Effects of Olfactory Stimulation in Patients with Severe Acquired Brain Injury
Brief Title: Olfactory Stimulation in Severe Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, PADUA LUCA, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4376
Record Dates: First submitted 2023-02-17; First posted 2023-02-28 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2024-02

CONDITIONS: Disorder of Consciousness
Keywords: Acquired Brain Injury; Disorder of Consciousness; Olfactory stimulation
MeSH Terms: conditions — Consciousness Disorders; Brain Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group natural_neutral_chemical (Experimental): The recruited subjects (DoC patients and healthy subjects) will be evaluated inside a quiet, well-ventilated room and will be subjected to olfactory stimulation using odors with different characteristics a "natural" type odor, e.g., mint, a "chemical" type odor, e.g., gasoline, and a "neutral" type odor, e.g., water.
  Stimulation will have, for each odor the duration of 5 minutes. It will always be carried out within the same time slot (between 8:00 am and 4:00 pm) for 5 consecutive days for 2 weeks. Before and after the administration of each odor, a neutral odor (water) will be administered as a control in the same manner as described above.
  The sequence of odor administration will be: natural odor (mint) for 5 minutes, neutral odor (water) for 5 minutes, chemical odor (gasoline) for 5 minutes.
  Interventions: Other: Olfactory sstimulation
- Group chemical:neutral_natural (Experimental): The recruited subjects (DoC patients and healthy subjects) will be evaluated inside a quiet, well-ventilated room and will be subjected to olfactory stimulation using odors with different characteristics a "natural" type odor, e.g., mint, a "chemical" type odor, e.g., gasoline, and a "neutral" type odor, e.g., water.
  Stimulation will have, for each odor the duration of 5 minutes. It will always be carried out within the same time slot (between 8:00 am and 4:00 pm) for 5 consecutive days for 2 weeks. Before and after the administration of each odor, a neutral odor (water) will be administered as a control in the same manner as described above.
  The sequence of odor administration will be: chemical odor (gasoline) for 5 minutes, neutral odor (water) for 5 minutes, natural odor (mint) for 5 minutes.
  Interventions: Other: Olfactory sstimulation

INTERVENTIONS:
Other: Olfactory sstimulation — The odors being tested (natural odor, neutral odor, chemical odor) are part of the 40 fragrances made by International Flavors and Fragrances (IFF) and each is contained in an approximately 15-mL glass bottle. The selected odors will be administered using a small paper strip (15 cm length and 0.7 cm width) that will be soaked in the selected odor and placed under the subject's nose at a minimum distance to prevent direct contact of the strip with the skin; the strip will be moved alternately from one nostril to the other.
  Stimulation will have, for each odor the duration of 5 minutes. It will always be carried out within the same time slot (between 8:00 am and 4:00 pm) for 5 consecutive days for 2 weeks. Before and after the administration of each odor, a neutral odor (water) will be administered as a control in the same manner as described above.
  The sequence of odor administration will be randomized according to a computer-generated sequence.

SUMMARY:
The management of patients with disorders of consciousness (DoC) represents a topic of great importance and topicality in the medical-scientific field because of the complexity and extent of associated disabilities and the difficulty in identifying effective therapeutic approaches. Despite significant advances in neuroscience, much remains to be elucidated about the mechanisms that regulate consciousness, and which of these to act on to stimulate plasticity and thus promote responsiveness and functional recovery in patients. Evidence on treatments that promote arousal and communication skills in individuals with DoC is still limited.

Among the possible interventions proposed in the literature, sensory stimulation would act by stimulating synaptic plasticity, counteracting the sensory deprivation to which these patients are exposed.

Published studies on the topic have produced results that are not unique and difficult to compare across different stimulation protocols (content, intensity, frequency, modality), settings and patient populations.

DETAILED DESCRIPTION:
Smell is a primitive and complex sense related to emotions, memory and language. When we smell an odor, its molecules reach the nasal cavity and bind to the receptors of olfactory neurons, which transform the chemical information into an electrical signal that reaches the olfactory bulb and is then transmitted to the brain areas (piriform cortex, amygdala, thalamus, hypothalamus, insula, anterior cingulate cortex, orbitofrontal cortex) deputed to the emotional perception of smell and its storage. Studies in the literature have demonstrated the ability of the olfactory stimulus to influence emotional and cognitive processes (attention, memory, language), motor gesture, and autonomic nervous system response in healthy subjects. The use of stimuli with emotional and familiar content for the subject has also been shown to increase the likelihood of observing a behavioral response in patients with DoC.

In DoC patients, the use of the olfactory stimulus (intensity, modality, timing, measurement tools) in the recovery process is still limited, and it has not yet been clarified what effect it has on awakening and neurovegetative nervous system response.

This study aims to investigate, in both healthy subjects and patients with obsessive compulsive disorder (DoC) resulting from severe Acquired Brain Injury (sABI), the effects that odors of various types produce at the level of the autonomic nervous system (ANS) and brain connectivity.

More specifically, this study aims to evaluate, in healthy subjects and in patients with DoC, the effects of neutral, pleasant, and unpleasant olfactory stimuli on ANS, brain connectivity, reactivity, and the possible onset of habituation following repeated administration of the same olfactory stimulus.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 90 years;
* Glasgow Come Scale (GCS) score between 8 and 13;
* Level of Cognitive Function (LCF) score between 2 and 3;
* Latency from the acute event of not more than 2 months;
* Spontaneous eye opening.

Exclusion Criteria:

* Documented history of brain injury prior to the one that resulted in hospitalization;
* Documented history of uncorrected visual or hearing impairment;
* Documented history of chronic rhinosinusitis with or without the presence of naso-sinus polyps;
* Previous history of psychiatric and/or neurological disorders that resulted in significant disability prior to the acute event;
* Acute pathology at the time of recruitment, head injury, or ischemic or expansive injury with suspected peripheral olfactory tract involvement.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Sympathetic Skin Response (SSR) | Change from baseline SSR at 2 weeks
  SSR is a physiologic measurement to record the electrical potential through an electrode placed on the palm of the hand after median nerve stimulation. The test is based on the temporary change in skin electrical resistance in response to activation of the sweat glands when exposed to a stimulus. It allows assessment of the ANS response through the study of sympathetic cholinergic efferent pathways

SECONDARY OUTCOMES:
Electrodermal Activity (EDA) | Change from baseline EDA at 2 weeks
  The E4 wereable medical devide (Empatica) will be used to assess the electrodermal activity (EDA).
  Fluctuations in some electrical properties of the skin will be recorded; the online software Empatica (https://www.empatica.com/en-eu/) will the export the recorded data.
  A higher EDA value corresponds to a higher stress level.
Heart Rate Variability (HRV) | Change from baseline HRV at 2 weeks
  HRV, that is, the assessment of heart rate variability, is evaluated using an electrocardiographic (ECG) device with normal surface electrodes applied at the level of the heart and special software for data analysis.
Electrocortical activity | Change from baseline EEG-HD at 2 weeks
  The information inherent in the assessment of electrocortical activity, will be recorded using 64-channel high density electroencephalogram (EEG-HD). The presence of a cortical potential in motor area will be assessed by following the somatotopic organization, by reconstructing a brain map in amplitude.
Coma Recovery Scale-revised | Change from baseline CRS-r at 2 weeks
  CRS-r is an assessment tool that examines 6 functions: auditory, visual, oral-verbal motor, communicative and vigilance.
  Its different items are organized hierarchically (low scores represent reflex activities, hig scores decribe cognitively mediated behaviours).
  For each function examined, the diagnosis of Vegetative State, Minimal Consciousness State, Emergence from Minimal Consciousness State can be made.

CONTACTS AND LOCATIONS:
Overall Officials: Luca Padua, MD, phD, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, RM, Italy